CLINICAL TRIAL: NCT03424343
Title: The Long-term Impact of Pediatric Cancer on Adolescents, Emerging Adults, and Their Family: Identity, Psychosocial Functioning, and Development
Brief Title: Longitudinal Identity Study of Childhood Cancer Survivors
Acronym: LInC
Status: Active, not recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Koen Luyckx, Associate professor at the Faculty of Psychology and Educational Sciences, KU Leuven
Other Study IDs: S60535
Record Dates: First submitted 2017-11-29; First posted 2018-02-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Cancer
Keywords: survivors; parents; sibling; family environment; psychosocial functioning; longitudinal; cancer; identity; adolescence; emerging adulthood
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer survivor, parents, sibling: study samples adolescent and young adult survivors of pediatric cancer, their parents, and one sibling; they are assessed using self-report questionnaires, so no intervention takes place
  Interventions: Other: Questionnaire bundle; Other: Obtaining information from survivors' medical file

INTERVENTIONS:
Other: Questionnaire bundle — Questionnaires on identity formation and psychosocial functioning, assessed and reported at baseline, one year later, two years later, and five years later.
Other: Obtaining information from survivors' medical file — After obtaining informed consent, we will access the medical file of participants to obtain information on the diagnosis, time of diagnosis, treatment duration, type of treatment, and relapse (when applicable).

SUMMARY:
The study investigators plan to conduct a longitudinal questionnaire study in adolescents and emerging adults (14-25 years of age at the start of the study) who survived childhood cancer to chart their identity development and broader social functioning. Additionally, the functioning of these survivors will be related to the functioning of their parents and siblings. The investigators shall focus especially on the current experience and impact of the earlier cancer experience. They will investigate to what extent the experience of a life-threatening disease has an effect on the daily life of survivors and over time and how the survivors develop through the course of adolescence and emerging adulthood on the psychosocial level. The formation of an adult identity is a very challenging task during adolescence and the way to adulthood and the fact that these youth had cancer during their childhood may especially complicate this process of identity formation. Furthermore, both parental and sibling functioning will be taken into account, which will allow us to examine inter-generational mechanisms (thus parental functioning that possibly impacts youth functioning and vice versa) and sibling functioning in these families. To investigate the latter, at each timepoint of the longitudinal study a sibling between 14 and 25 years of age at the start of the study will be included (if there is more than one sibling in a family, ideally the sibling who is closest in age will be the one who participates in the study). Moreover, a community sample that is matched on age and sex with the survivor of pediatric cancer will be assessed. This will allow the investigators to make well-founded comparisons regarding identity development and broader psychosocial functioning.

DETAILED DESCRIPTION:
In the present longitudinal study, four main research questions will be investigated.

1. How does identity develop in cancer survivors? Based on previous findings from studies in identity development, it seems that young adults with a chronic disease like type 1 diabetes show less exploration or consider less identity possibilities from which they can choose, e.g. they dwell less upon the choice of education. Does this finding also apply to survivors of childhood cancer or are these youth more similar to a community sample? This research question may provide an answer to the question whether or not there is a continued (psychological) impact of childhood cancer on the later identity development of survivors. For this purpose the investigators shall make use of an identity model which was developed at their research department and which has gained much international research attention. In addition, the investigators want to look at illness-identity, which comprises the amount to which the earlier cancer experience is integrated into one's identity. Does the youngster feel still engulfed by the earlier cancer experience, or has he/she integrated this experience as part of his/her self-concept? Or does the youngster feel even enriched by the earlier cancer experience, thus did he/she end up even stronger through the experience?
2. How do survivors of pediatric cancer and/or their parents function on the psychological level, more specific on the level of life satisfaction and depressive symptoms, and what is the role of identity and personality variables herein? This question examines, among other factors, concepts like benefit-finding, post-traumatic growth, resilience,... Thereby it would be interesting to examine whether different subgroups can be identified, for example, which groups of persons display less adaptive functioning and why?
3. Are there certain parenting dimensions (e.g. overprotection, responsiveness, psychological control,...) which are more prevalent in families that were confronted with pediatric cancer and are these dimensions differently related to the psychosocial adaptation of survivors? Does this relate to certain aspects of survivor functioning, like depressive symptoms and quality of life? Thereby, transactional processes between survivor and parental functioning will be investigated, e.g. does identity development of survivors have an impact on parental well-being, and has parental well-being in turn an impact on survivor functioning? Taken together, the investigators want to investigate to what extent these contextual variables determine the functioning of adolescents and emerging adults.
4. What is the impact for siblings of cancer survivors? How do they go through their identity process? Do they experience the same parenting as the survivors experience themselves? E.g if survivors would experience more parental overprotection, would siblings experience overprotection to the same extent?

ELIGIBILITY:
Inclusion Criteria:

* Survivors of childhood leukemia/lymphoma, solid tumors, and brain tumors, of whom the treatment has ended.
* 14-25 years at the start of the study
* Treated at the department of pediatric oncology at University Hospital Leuven, Belgium.
* Sufficient knowledge of Dutch

Exclusion Criteria:

* Mental retardation which hinders completion of the questionnaire bundle
* Younger than 14 year and older than 25 year
* Physically incapable to complete the questionnaire bundle
* Insufficient knowledge of Dutch
* Contact information is not available

Ages: 14 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Survivors of childhood cancer, treated at the department of pediatric oncology at UZ Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Dimensions of Identity Development | Assessed and reported at baseline, one year later, two years later, and five years later
  Dimensions of Identity Development Scale (DIDS); dimensions: commitment making (range: 5 - 25), Identification with Commitment (range: 5 - 25), Exploration in Breadth (rang: 5 - 25), Exploration in Depth (range: 5 - 25), Ruminative Exploration (range: 5 - 25); for each dimension, a higher score indicates more identification with the dimension
Change in Identity from an Eriksonian Perspective | Assessed and reported at baseline, one year later, two years later, and five years later
  Erikson Psychosocial Stage Inventory (EPSI); subscales: Synthesis (range: 5 - 30), Confusion (range: 5 - 30); for each scale, higher scores indicate more identification with the scale
Change in Illness Centrality | Assessed and reported at baseline, one year later, two years later, and five years later
  Illness Centrality; total scale range: 0 - 4; A higher score indicates more identification with the scale
Change in Self-Identity after Cancer | Assessed and reported at baseline, one year later, two years later, and five years later
  Self-Identity after Cancer; dimensions: victim of cancer (range: 1 - 5), cancer patient (range: 1 - 5), person who had cancer (range: 1 - 5), survivor (range: 1 - 5); for each dimension, a higher score indicates more identification with the dimension

SECONDARY OUTCOMES:
Change in Post-Traumatic Stress Symptoms (measured in survivors) | Assessed and reported at baseline, one year later, two years later, and five years later
  Children's Revised Impact of Event Scale (CRIES-13); total scale range: 0 - 65; Higher scores indicate more sensitivity for PTSD; A score higher than 30 possibly indicates the presence of PTSD; subscales: Intrusion (range: 0 - 20), Avoidance (range: 0 - 20), Arousal (range: 0 - 25); Higher scores indicate more identification with the scale
Change in Illness-related Benefit Finding (measured in survivors) | Assessed and reported at baseline, one year later, two years later, and five years later
  Benefit scale from the Benefit and Burden Scale (BBSC); total scale range: 10 - 50; A higher score indicates more identification with the scale
Change in Depressive Symptoms (measured in survivors, siblings, and parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Center for Epidemiologic Studies Depression (CES-D-12); total scale range: 0 - 36; a higher score indicates the presence of more depressive symptoms
Change in Cancer-related Worries (measured in survivors and parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Cancer Related Worries Scale; total scale range: 4 - 20; A higher score indicates the presence of more cancer-related worries
Change in Global Life Satisfaction (measured in survivors, siblings and parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Satisfaction with Life Scale (SWLS); total scale range: 5 - 35; A higher score indicates more satisfaction with life
Change in Bodily Functioning (measured in survivors) | Assessed and reported at baseline, one year later, two years later, and five years later
  Short Form 36, physical subscale (SF-36); total scale range: 10 - 30: A higher score indicates worse bodily functioning
Change in Self-Esteem (measured in survivors, siblings, and parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Rosenberg Self-Esteem Scale (RSES); total scale range: 10 - 40: A higher score indicates higher self-esteem
Change in Resilience (measured in survivors and parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Brief Resilience Scale (BRS); total scale range: 6 - 30; A higher score corresponds to being more resilient
Change in Personality (measured in survivors and siblings) | Assessed and reported at baseline, one year later, two years later, and five years later
  Big Five Inventory 10 (BFI-10); subscales: Extraversion (range: 2 - 10), Agreeableness (range: 2 - 10), Conscientiousness (range: 2 - 10), Neuroticism (range: 2 - 10), Openness (range: 2 - 10); for each scale, a higher score indicates more identification with the scale
Change in Self-Harm (measured in survivors) | Assessed and reported at baseline, one year later, two years later, and five years later
  Based on Goossens et al., 2013: Health risk behaviors in adolescents and emerging adults with congenital heart disease: psychometric properties of the Health Behavior Scale-Congenital Heart Disease
Change in Perception of Control (measured in survivors, siblings, and parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Multidimensional Health Locus of Control Scale (MHLCS): subscales: Internal Health Locus of Control (range 6 - 36), Powerful Others Health Locus of Control (range 6 - 36), Chance Health Locus of Control (range: 6 - 36); for each scale, a higher score indicates more identification with the scale
Change in Social Support (measured in survivors and siblings) | Assessed and reported at baseline, one year later, two years later, and five years later
  Multidimensional Scale of Perceived Social Support (MSPSS); subscales: support from special someone (range: 4 - 28), support from family (range: 4 - 28), support from friends (range: 4 - 28); for each subscale, a higher score indicates more support
Change in Contact with Peer Survivors (measured in survivors) | Assessed and reported at baseline, one year later, two years later, and five years later
  Self-constructed questionnaire
Change in Parental Behavioral Control (measured in survivors, parents, and siblings) | Assessed and reported at baseline, one year later, two years later, and five years later
  Based on the 8-item Parental Expectations for Behavior Scale and the 8-item Parental Monitoring of Behavior Scale uit de 'Parental Regulation Scale - Youth Self-Report' (PRS -YSR; Barber, 2002); Behavioral Control; total scale range: 7 - 35; A higher score indicates more parental behavioral control
Change in Parental Responsiveness (measured in survivors, parents, and siblings) | Assessed and reported at baseline, one year later, two years later, and five years later
  Child Report of Parent Behavior Inventory (CRPBI; Schaefer, 1965; Schludermann & Schludermann, 1988); Responsiveness; total scale range: 7 - 35; A higher score indicates more parental responsiveness
Change in Parental Overprotection (measured in survivors, parents, and siblings) | Assessed and reported at baseline, one year later, two years later, and five years later
  based on Dutch Multidimensional Overprotective Parenting Scale, Kins & Soenens, 2013; Overprotection / anxious parenting; Overprotection; total scale range: 8 - 40; A higher score indicates more parental overprotection
Change in Parental Psychological Control (measured in survivors, parents, and siblings) | Assessed and reported at baseline, one year later, two years later, and five years later
  8-item Psychological Control Scale-Youth Self-Report ( Barber, 1996); Psychological Control; total scale range: 8 - 40; A higher score indicates more parental psychological control
Change in Illness Intrusiveness (measured in parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Illness Intrusiveness Questionnaire Parent Report (IIQ-Parent Report); total scale range: 13 - 91; A higher score indicates more illness intrusiveness
Change in Parental competence (measured in parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Parenting Stress Index - Sense of Competence Scale; total scale range: 13 - 78; A higher score indicates a lower sense of parental competence
Change in Role Restriction (measured in parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Parental Burden Questionnaire, subscale role restriction; total scale range: 6 - 24; A higher score indicates a greater sense of role restriction
Change in Relationship Quality (measured in parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Family Functioning Questionnaire, subscale parental relationship quality; total scale range: 5 - 20; A higher score indicates a greater sense of partner relationship quality
Change in Benefit Finding (measured in parents) | Assessed and reported at baseline, one year later, two years later, and five years later
  Benefit Finding Scale; total scale range: 15 - 105; A higher score indicates more benefit finding

CONTACTS AND LOCATIONS:
Overall Officials: Koen Luyckx, Dr., Principal Investigator — KU Leuven
Locations (1):
- Gasthuisberg, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No